CLINICAL TRIAL: NCT04298476
Title: Defining the Optimal Location to Place Local Anesthetic for an Adductor Canal Block for Pediatric Knee Arthroscopy Patients
Brief Title: Defining the Optimal Location to Place an Adductor Canal Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Aysha Hasan, Pediatric Anesthesiologist, Drexel University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1901006926
Record Dates: First submitted 2020-02-18; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- A (Placebo Comparator): Saline will be placed in syringe instead of ropivicaine 0.2% and the nerve block will be placed in the adductor canal at the desired location by the anesthesiologist
  Interventions: Procedure: Placement of an adductor canal nerve block
- B (Active Comparator): An adductor canal block will be placed with local anesthetic in the proximal 1/3 of the operative leg
  Interventions: Procedure: Placement of an adductor canal nerve block
- C (Active Comparator): An adductor canal block will be placed with local anesthetic in the middle 1/3 of the operative leg
  Interventions: Procedure: Placement of an adductor canal nerve block
- D (Active Comparator): An adductor canal block will be placed with local anesthetic in the distal 1/3 of the operative leg
  Interventions: Procedure: Placement of an adductor canal nerve block

INTERVENTIONS:
Procedure: Placement of an adductor canal nerve block — An adductor canal nerve block will be placed in a patient undergoing a knee arthroscopy in 1 of 3 locations with local anesthetic or placebo (without location definition or local anesthetic) to assess optimal placement of local anesthetic, pain management and anxiety scores post operatively.

SUMMARY:
The aim of the current project is to address a gap in the existing literature related to optimal placement of local anesthetic for an adductor canal (AC) block. The current study seeks to examine whether placement of the local anesthetic in the AC for knee surgery is more effective at reducing post-operative pain following arthroscopic knee surgery compared to a control. Specifically, if the anesthetic is more beneficial than the control group, the research will determine which location is optimal by comparing groups that receive anesthetic in the midpoint of the thigh, the proximal end of the thigh, or the distal end of the thigh.

DETAILED DESCRIPTION:
Although there has been an abundance of literature highlighting the efficacy of using regional blocks to decrease post-operative pain, the exact location of placement of local anesthetic for anesthetizing the nerves in the AC is unknown for optimal pain relief in patients undergoing knee surgery. The saphenous nerve consistently lies in the AC at various points of local anesthetic deposit, however there are many other nerves that lie in the canal that may branch off proximally or distally from the AC that are important to target in achieving optimal pain relief for patients undergoing knee arthroscopy.1-3 The AC is bounded in a triangular shape by the vastus medialis anterolaterally, the sartorius medially, and the adductor longus/adductor magnus posteriorly. The canal contains the deep femoral artery and the deep femoral vein. The saphenous nerve consistently lies within this canal, a significant sensory contributor to the knee.1-3 Other branches of the femoral nerve can also be found in the AC. The nerve to the vastus medialis (NVM) and the posterior branches of the obtruator nerve (PON) can also be found, although inconsistently, in the AC at various locations.4,5 These nerves are thought to innervate the knee as well and contribute to pain when missed during this block. The course of these nerves is unknown. While some surmise that the NVM branches proximally and the PON branches distally, there is no consensus on this.

Currently, an AC block is most often placed in the mid-thigh as measured by visual observation. The investigators seek to investigate where along the tract of the AC would be optimal to place local anesthetic to optimize analgesia on all nerves that innervate the knee without having motor loss as would occur with a femoral nerve block

ELIGIBILITY:
Inclusion Criteria:

* Patient is 7 to ≤ 17 years of age
* Patient at St. Christopher's Hospital for Children
* Receiving a knee arthroscopy procedure
* English speaking

Exclusion Criteria:

* Patient is less than 7 years of age or over 17 years of age
* Patient has cognitive impairments
* Patient had previous operations on the same lower extremity as the current knee arthroscopy
* Patient has a positive B-HCG (identified through urine or blood test)
* Patient does not speak English

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Reported pain as assessed by Wong-Baker FACES scale | 48 hours
  Patient self-reported pain intensity following the procedure. The scale ranges from 0-10 (0 = no pain; 10 = extreme). Collected at two points: pre-and-post procedure.

SECONDARY OUTCOMES:
Patient reported anxiety as assessed by the Child's Anxiety Meter-State (CAM-S) | 48 hours
  Patient self-reported anxiety levels will be measured on a thermometer-style graphic, where the bottom (near the base) represents low anxiety and the top represents high levels of anxiety.
Parent reported anxiety as assessed by the Child's Anxiety Meter-State (CAM-S | 48 hours
  Parent self-reported anxiety levels will be measured on a thermometer-style graphic, where the bottom (near the base) represents low anxiety and the top represents high levels of anxiety
Patient reported sensation through ice and pinprick | 48 hours
  Patients will report sensation on their knee postoperatively by reponding if they can (yes) or cannot (no) feel a pinprick and piece of ice.
Usage of narcotic pain medication | 48 hours
  The amount of narcotic pain medication that the patients utilize after their discharge will be documented as morphine milligram equivalents (e.g., MME).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong WY, Bjorn S, Strid JM, Borglum J, Bendtsen TF. Defining the Location of the Adductor Canal Using Ultrasound. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):241-245. doi: 10.1097/AAP.0000000000000539. PMID 28002228
- [Background] Bendtsen T.F., Lopez A.M., Clark T.B. (2018). Ultrasound-Guided Saphenous (Subsartorius/Adductor Canal) Nerve Block. NYSORA Continuing Medical Education. Retrieved from https://www.nysora.com/ultrasound-guided-saphenous-subsartoriusadductor-canal-nerve-block
- [Background] Burckett-St Laurant D, Peng P, Giron Arango L, Niazi AU, Chan VW, Agur A, Perlas A. The Nerves of the Adductor Canal and the Innervation of the Knee: An Anatomic Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):321-7. doi: 10.1097/AAP.0000000000000389. PMID 27015545
- [Background] Quemby D. & McEwen A. (2014). Ultrasound Guided Adductor Canal Block (Saphenous Nerve Block). Anesthesia Tutorial of the Week. Retrieved from https://www.aagbi.org/sites/default/files/301%20Ultrasound%20Guided%20Adductor%20Canal%20(Saphenous%20Nerve)%20Block.pdf
- [Background] Runge C, Moriggl B, Borglum J, Bendtsen TF. The Spread of Ultrasound-Guided Injectate From the Adductor Canal to the Genicular Branch of the Posterior Obturator Nerve and the Popliteal Plexus: A Cadaveric Study. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):725-730. doi: 10.1097/AAP.0000000000000675. PMID 28937534
- [Background] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126